CLINICAL TRIAL: NCT03191929
Title: Depression Screening in Primary Care: Using HIT for Patients With Limited English
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dara Sorkin (Other)
Responsible Party: Sponsor-Investigator, Dara Sorkin, Associate Professor, University of California, Irvine
Organization: University of California, Irvine (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2011-8343
Record Dates: First submitted 2017-06-09; First posted 2017-06-19 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Depression; Post-Traumatic Stress Disorder
Keywords: Depression; Post-traumatic Stress Disorder; Health Information Technology (HIT); Primary Care Provider; Mental Health Screening
MeSH Terms: conditions — Depression; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HIT Intervention Arm (Experimental): The Health Information Technology Intervention Study Arm consisted of: 1) web-based tutorial on delivering trauma-informed care, 2) Multi-media mental health risk assessment, 3) Immediate provider notification, which included flagging patients' scores that met criteria for symptoms of depression and/or PTSD, 4) subsequent integration into the patient electronic medical record, and 5) Clinical decision support adapted from the Harvard Program in Refugee Trauma.
  Interventions: Other: HIT Intervention
- Minimal Intervention Control Arm (Active Comparator): The Minimal Intervention Control Arm consisted of: 1) web-based tutorial on delivering culturally competent health care in general, 2) Multi-media mental health risk assessment, 3) Provider notification only in the event that patients' scores evidenced symptoms of being at risk to harm either themselves or others.
  Interventions: Other: Minimal Intervention Control Arm

INTERVENTIONS:
Other: HIT Intervention — Patients in the HIT intervention completed a multi-media, culturally adapted, mental health risk assessment tool in their preferred language prior to their baseline health care visit with their primary care provider. Patients' scores were transmitted to the provider prior to their clinic visit.
  Providers in the HIT intervention received a web-based training developed by the Harvard Program in Refugee Trauma to train providers in delivering culturally competent, trauma-informed care to address mental health problems and other trauma-related medical issues in patients who experienced extreme war trauma. Providers also received ongoing clinical decision support through a mobile application to support the diagnosis and initiation of treatment for depression and/or PTSD.
  Arms: HIT Intervention Arm
Other: Minimal Intervention Control Arm — Patients in the Minimal Intervention Control Arm completed a multi-media, culturally adapted, mental health risk assessment tool in their preferred language prior to their baseline health care visit with their primary care provider; however, patients' scores in the Minimal Intervention Control Arm were only transmitted to the provider prior to their clinic visit if they showed evidence of being at risk to harm either themselves or others.
  Providers in the Minimal Intervention Control Arm completed the online tutorial, "A physician's practical guide to culturally competent care," which was provided by The Office of Minority Health, US Department of Health and Human Services Website.
  Arms: Minimal Intervention Control Arm

SUMMARY:
This study assessed the potential of Health Information Technology (HIT) to improve the screening, diagnosis, and treatment of depression and post-traumatic stress among LEP Southeast Asians. Should this intervention be found to be effective, the principles of the HIT technology could be easily adapted for screening in other languages to increase the recognition and treatment of depression and PTSD in primary care settings.

DETAILED DESCRIPTION:
The prevalence of depression in primary care is high. Primary care physicians serve as the initial point of contact for most patients with depression, yet it is estimated that only about half of the depressed patients who present for care are recognized and treated. Language barriers can further exacerbate this problem. Approximately 54 million people in the United States speak a language other than English at home and over 21 million are limited English-language proficient (LEP). Language barriers may result in less discussion about patients' mental health needs and fewer referrals to specialty mental health services. Recent advances in health information technology (HIT), however, may facilitate novel ways to screen for mental health problems among limited English proficient patients. The HIT intervention is a provider-level intervention that consists of four components: 1) web- based training for the providers; 2) multimedia electronic screening of patients for depression and PTSD; 3) immediate notification to the health care providers and integration with the patients' electronic health records (EHR); and 4) provider clinical decision support. In a randomized controlled trial in a primary care setting, we will assess the potential of a multi-component health information technology intervention to improve the screening rates, clinical detection, provider initiation of treatment, and patient outcomes for depression and post-traumatic stress disorder among LEP Southeast Asians. We will examine the usability and acceptability of this technology to patients with limited English skills and their providers. Finally, we will identify and evaluate potential facilitators and barriers to wide spread implementation and dissemination of the HIT intervention. This technology has the potential to be adapted and utilized for any group of limited English-language proficient (LEP) patients, regardless of their native language, and has the potential to be adapted for providers to aid in the recognition, diagnosis, and treatment of mental health problems in diverse primary care settings.

ELIGIBILITY:
Inclusion Criteria:

* Cambodian patients over age 18 were included.

Exclusion Criteria:

* Patients with severe visual/hearing impairments, major psychiatric disorders such as bipolar disorder or schizophrenia, and/or life-threatening illness, which limited their ability to consent to the study were excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 410 (Actual)
Dates: Start 2011-08; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Appropriate clinical detection of depression and/or PTSD | 12 weeks
  The appropriate presence or absence of provider diagnosis of depression and/or PTSD in the patient electronic medical record.

SECONDARY OUTCOMES:
Provider initiation of guideline mental health treatment and trauma informed care | 12 weeks
  The study will examine whether providers in the HIT intervention group were more likely to initiate guideline mental health treatment and trauma-informed care relative to the control group. The initiation of guideline mental health treatment and trauma-informed care will be examined by obtaining providers' documentation and treatment plans for each patient's clinic visits over 12 weeks. Providers will receive credit for initiating guideline mental health treatment if they initiated one or more of the following recommendations: 1) Pharmacotherapy discussion and prescription, 2) watchful waiting, and 3) referral to mental health specialist. Providers will receive credit for initiating trauma-informed care if the provider engaged in one or more of the following: 1) conducted a risk assessment of patients' depression or PTSD status, 2) discussed the trauma story with the patient, 3) asked patients if they wanted to improve their well-being, and/or 4) assessed psychiatric symptoms.
Patient outcomes (at 12 weeks post-baseline visit) for depression and/or PTSD | 12 weeks
  The study will examine whether patients' self-reported outcomes (12 weeks post-baseline visit) for depression and/or PTSD will be improved by the HIT intervention. Depression and PTSD status will be assessed by the HSC and HTQ, which was readministered at 12 weeks post-baseline.
Patients' evaluation of the overall quality of care | 12 weeks
  Patients' evaluation of their overall quality of care will be assessed using a single item that asked them to rate the quality of care they received in the past 12 months. Ratings were made on a 5-point scale (1 = Poor, 5 = Excellent).
Patients' level of involvement in decision-making related to their care | 12 weeks
  Patients' level of involvement in decision-making related to their care will be assessed using the Participatory Decision Making Scale (PDM-7). Ratings were made on a 5-point Likert scale (1=Never/None of the time; 5=Very often/All of the time). A sample item included "How often do the doctors that take care of you offer you choices in your medical care?"
Patients' trust in their provider | 12 weeks
  Patients' trust in their provider will be assessed using five items from the Trust in Physicians Scale. Ratings were made on a 5-point Likert scale (1=Never, 5=Always). A sample item included "How often do you feel you trust your doctor's judgments about your medical care?"
Patients' perceptions of being treated as an equal partner in their care | 12 weeks
  Patients' perceptions of being treated as an equal partner by their provider will be assessed by a single item, "Do the doctors who care for you make an effort to treat you like an equal partner?" Ratings were made on a 5-point scale (1=Definitely Yes; 5=Definitely No)

CONTACTS AND LOCATIONS:
Overall Officials: Dara H. Sorkin, Ph.D., Principal Investigator — University of California, Irvine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sorkin DH, Rizzo S, Biegler K, Sim SE, Nicholas E, Chandler M, Ngo-Metzger Q, Paigne K, Nguyen DV, Mollica R. Novel Health Information Technology to Aid Provider Recognition and Treatment of Major Depressive Disorder and Posttraumatic Stress Disorder in Primary Care. Med Care. 2019 Jun;57 Suppl 6 Suppl 2(Suppl 6 2):S190-S196. doi: 10.1097/MLR.0000000000001036. PMID 31095060